CLINICAL TRIAL: NCT04242992
Title: Testing the Effectiveness of an Evidence-based Transdiagnostic Cognitive Behavioral Therapy Approach for Improving HIV Treatment Outcomes Among Violence-affected and Virally Unsuppressed Women in South Africa
Brief Title: Effectiveness of Transdiagnostic Cognitive Behavioral Therapy for Improving HIV Treatment Outcomes in South Africa
Acronym: CETA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-39746; 1R01MH121998 (NIH)
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: HIV/AIDS; Violence
Keywords: HIV; Retention; Viral suppression; Violence; Cognitive behavioral therapy (CBT); Common Elements Treatment Approach (CETA)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Spermine Synthase

STUDY DESIGN:
Intervention Model Description: Women will be randomized 1:1 to either CETA or an active attention control arm.
Who Masked: Outcomes Assessor
Masking Description: As the intervention is a behavioral intervention, it will not be possible to blind women to their intervention, but outcome assessors will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CETA (Common Elements Treatment Approach) (Experimental): CETA is a modular, multi-problem, flexible psychotherapy approach that trains a lay provider in nine evidence-based cognitive behavioral therapy (CBT) elements so the provider can treat a variety of common problems, including violence, substance use, depression, anxiety, risky behaviors (sexual, non-adherence), and other trauma-related symptoms. Patients randomized to CETA will meet weekly with a lay provider or community health worker member of the study staff for about an hour once each week, approximately 6-12 times depending on presentation and symptom level. This treatment arm will include Short Message Service (SMS) text reminders of their HIV care appointments, similar to the active control group. As of October 12, 2022 participants can elect to have CETA delivered by telephone.
  Interventions: Behavioral: CETA; Other: Short Message Service (SMS) text reminders
- Active control (Active Comparator): Our comparison arm will be an active control receiving usual care for intimate partner violence. Short Message Service (SMS) text messages will be sent monthly to our control group participants to remind them of HIV care appointments.
  Interventions: Other: Short Message Service (SMS) text reminders

INTERVENTIONS:
Behavioral: CETA — CETA is a modular, multi-problem, flexible psychotherapy approach that trains a lay provider in nine evidence-based CBT elements so providers can treat a variety of common problems, including violence, substance use, depression, anxiety, risky behaviors (sexual, non-adherence), and other trauma-related symptoms. Patients randomized to CETA will meet weekly with a lay provider or community health worker member of the study staff for about an hour once each week, approximately 6-12 times depending on presentation and symptom level. This treatment arm will include SMS reminders of their HIV care appointments, similar to the active control group.
  Arms: CETA (Common Elements Treatment Approach)
Other: Short Message Service (SMS) text reminders — Short Message Service (SMS) text reminders for upcoming appointments will be sent monthly.

SUMMARY:
This study will evaluate the impact of the Common Elements Treatment Approach (CETA), an evidence-based intervention comprised of cognitive-behavioral therapy elements, at improving HIV treatment outcomes among women with HIV who have experienced intimate partner violence (IPV) and have an unsuppressed viral load on HIV treatment. To evaluate CETA, the investigators will conduct a randomized controlled trial of HIV-infected women, with or without their partners, who have experienced IPV and have an unsuppressed viral load to test the effect of CETA in increasing viral suppression and reducing violence. The investigators will also identify mediators and moderators of CETA's effect on retention and viral suppression and assess the cost and cost-effectiveness of CETA vs. active control at increasing the proportion who are retained and virally suppressed by 12 months.

DETAILED DESCRIPTION:
There are just under one million people with HIV in South Africa who have initiated antiretroviral therapy (ART) but remain unsuppressed. South Africa has been making progress towards UNAIDS 90-90-90 targets but currently only 47% of those infected are suppressed. In South Africa, one major barrier to consistent treatment is intimate partner violence (IPV); nearly 50% of women have experienced IPV. The Common Elements Treatment Approach (CETA) is an evidence-based intervention intended to provide coping skills to women who have experienced IPV, and is comprised of cognitive-behavioral therapy elements. It is a transdiagnostic tool that can flexibly address a range of mental health problems (e.g. depression, anxiety) and represents the current best practice in global mental health as a more cost-effective, scalable and sustainable model. CETA is one of the most promising interventions to impact HIV outcomes through addressing the indirect effects of IPV on adherence and continuity of care.

The investigators will conduct a randomized controlled trial of HIV-infected women, with or without their partners, who have experienced IPV and have an unsuppressed viral load to test the effect of CETA, in increasing retention and viral suppression, and reducing violence. The study has three aims:

* Aim 1: Among HIV-infected women on ART who have experienced IPV and have an unsuppressed viral load, assess the effectiveness of CETA vs. active control at increasing the proportion retained and virally suppressed by 12 months and at decreasing the severity and incidence of IPV and other mental and behavioral health problems using an individually randomized trial;
* Aim 2: To identify mediators and moderators of CETA's effect on the primary outcome (retention and viral suppression);
* Aim 3: To assess the cost and cost-effectiveness of CETA vs. active control at increasing the proportion who are retained and virally suppressed by 12 months.

Study staff will obtain full informed consent from those who meet inclusion criteria. For those that agree to participate, study staff will then randomize patients to CETA or control using sealed randomization envelopes. All subjects will be followed for 24 months to ensure data for primary and secondary outcomes is complete. Follow-up HIV data will be passive using routinely collected medical records from the clinics. HIV outcomes will be assessed at 3-, 12- and 24-months post-baseline. Questionnaires on violence, substance use, and mental health will be administered at baseline, and at 3 months (following CETA end) and 12 months post-baseline. These include: Severity of Violence Against Women Scale, Center for Epidemiological Studies-Depression Scale, Harvard Trauma Questionnaire, and Alcohol, Smoking, and Substance Involvement Screening Test. The primary outcome will be retention and viral suppression (<50 copies/mL) by 12 months after randomization. Secondary outcomes will include: 1) Viral suppression at 3 and 24 months; 2) Attrition at 12 and 24 months; 3) IPV, mental/behavioral health, alcohol and other substance use at 3 and 12 months; and 4) Cost and cost-effectiveness of the intervention.

The primary aim is to analyze the impact of CETA in the full study population; however, our sample size was calculated to ensure our ability to detect differences separately among women who include a partner in the CETA intervention and those who do not. A sample of 400 women will be included which will give us 80% power to detect an absolute 21% difference between arms. The primary analysis will be a comparison of intervention and control by risk differences with 95% confidence intervals. The investigators will analyze direct effects of CETA on continuous outcomes (e.g., mental health) with linear mixed models.The impact of potential moderators on retention and mental health outcomes using interaction terms will be assessed. Micro costing methods will be used to cost all resources utilized and the cost effectiveness of CETA achieving the primary outcome will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult HIV positive women
* Initiated HIV treatment
* Most recent viral load >50 copies/mL or they have defaulted from treatment or had a missed or late (>14 days) visit in the last year
* Has experienced IPV in the past 12 months
* Has their own phone and can receive text messages
* Literate and able to speak and read one of: English, Zulu, SeSotho
* If including a partner, the woman has disclosed HIV status to the partner that will be invited to participate

Exclusion Criteria:

* Unwilling to complete the informed consent process
* Currently psychotic or on unstable psychiatric regimen
* Suicide attempt/ideation with intent and plan, and/or self-harm in the past month
* Enrolled in any other HIV treatment intervention study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
12 month viral suppression | 12 months post randomization
  The proportion of participants who are virally suppressed (<50 copies/mL) by 12 months post randomization

SECONDARY OUTCOMES:
3 month viral suppression | 3 months post randomization
  The proportion of participants who are virally suppressed (<50 copies/mL) by 3 months post randomization
24 month viral suppression | 24 months post randomization
  The proportion of participants who are virally suppressed (<50 copies/mL) by 24 months post randomization
12 month attrition rate | 12 months post randomization
  Attrition rate (the opposite of retention) will be defined as the proportion of participants being more than 90 days late for a study visit 12 months post randomization.
24 month attrition rate | 24 months post randomization
  Attrition rate (the opposite of retention) will be defined as the proportion of participants being more than 90 days late for a study visit 24 months post randomization.
Change in violence against women from baseline to 3 months | Baseline to 3 months
  Violence will be measured using the Severity of Violence Against Women Scale (SVAWS) physical/sexual violence subscale, a 27 item measure with a possible range of 27-108 and higher scores associated with greater severity of experienced violence.
Change in violence against women from baseline to 12 months | Baseline to 12 months
  Violence will be measured using the Severity of Violence Against Women Scale (SVAWS) physical/sexual violence subscale, a 27 item measure with a possible range of 27-108 and higher scores associated with greater severity of experienced violence.
Change in substance use from baseline to 3 months | Baseline to 3 months
  Substance use will be measured with the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST), which includes 7 items on frequency of use, abuse, and dependence symptoms for the following substance types: tobacco, alcohol, inhalants, marijuana, cocaine, amphetamines, sedatives, hallucinogens, opioids , or other substance. Higher scores are associated with greater substance involvement.
Change in substance use from baseline to 12 months | Baseline to 12 months
  Substance use will be measured with the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST), which includes 7 items on frequency of use, abuse, and dependence symptoms for the following substance types: tobacco, alcohol, inhalants, marijuana, cocaine, amphetamines, sedatives, hallucinogens, opioids , or other substance. Higher scores are associated with greater substance involvement.
Change in post-traumatic stress disorder (PTSD) symptoms from baseline to 3 months | Baseline to 3 months
  PTSD symptoms will be assessed using 16 items scored on a four-point scale (1 = none, 2 = some of the time, 3 = a lot of the time, 4 = most of the time) from the Harvard Trauma Questionnaire (HTQ). Higher scores are associated with greater PTSD symptom severity.
Change in post-traumatic stress disorder (PTSD) symptoms from baseline to 12 months | Baseline to 12 months
  PTSD symptoms will be assessed using 16 items scored on a four-point scale (1 = none, 2 = some of the time, 3 = a lot of the time, 4 = most of the time) from the Harvard Trauma Questionnaire (HTQ). Higher scores are associated with greater PTSD symptom severity.
Change in Center for Epidemiological Studies-Depression Scale (CES-D) scale score from baseline to 3 months | Baseline to 3 months
  CES-D is a 20-item scale of depression with a possible range of 0-60 (total scale score). Higher scores are associated with greater depression symptom severity.
Change in Center for Epidemiological Studies-Depression Scale (CES-D) scale score from baseline to 12 months | Baseline to 12 months
  CES-D is a 20-item scale of depression with a possible range of 0-60 (total scale score). Higher scores are associated with greater depression symptom severity.
Cost-effectiveness | 12 months
  The incremental cost-effectiveness of CETA versus active control will be estimated for achieving the primary study outcome, retained in care and virally suppressed by 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Fox, DSc, Principal Investigator — Boston University
Locations (1):
- HIV Clinic, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Once the research team has had sufficient time to analyze the data and submit the results for the primary study aims, the data will be made available on request in de-identified format.
Supporting Information: Study Protocol, SAP
Time Frame: Once the primary aims are completed, approximately 12 months after study completion.

REFERENCES:
- [Derived] Zheng A, Kane JC, Mngadi-Ncube S, Fox MP, Manganye P, Long L, Metz K, Sardana S, Alto M, Greener R, Thea DM, Murray LK, Pascoe S. Effectiveness of the Common Elements Treatment Approach for mental and behavioural health outcomes among women struggling to remain adherent to HIV treatment and who have experienced intimate partner violence in South Africa: secondary outcomes from a randomised controlled trial. BMJ Ment Health. 2026 Jan 27;29(1):e302246. doi: 10.1136/bmjment-2025-302246. PMID 41592903
- [Derived] Zheng A, Kane JC, Mngadi-Ncube S, Fox MP, Manganye P, Long L, Metz K, Sardana S, Alto M, Greener R, Thea DM, Murray LK, Pascoe S. Effectiveness of the Common Elements Treatment Approach (CETA) for mental and behavioral health outcomes among women struggling to remain adherent to HIV treatment and who have experienced intimate partner violence in South Africa: A randomised controlled trial. medRxiv [Preprint]. 2025 Oct 15:2025.10.14.25337970. doi: 10.1101/2025.10.14.25337970. PMID 41282709
- [Derived] Pascoe S, Fox M, Kane J, Mngadi S, Manganye P, Long LC, Metz K, Allen T, Sardana S, Greener R, Zheng A, Thea DM, Murray LK. Study protocol: A randomised trial of the effectiveness of the Common Elements Treatment Approach (CETA) for improving HIV treatment outcomes among women experiencing intimate partner violence in South Africa. BMJ Open. 2022 Dec 22;12(12):e065848. doi: 10.1136/bmjopen-2022-065848. PMID 36549749